CLINICAL TRIAL: NCT06502652
Title: Effects of Hippo Therapy Versus Balance Training on Balance and Functional Mobility in Children With Down's Syndrome
Brief Title: Hippotherapy Versus Balance Therapy on Funvtional Mobility in Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0797
Record Dates: First submitted 2024-06-11; First posted 2024-07-16 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Down Syndrome
Keywords: Balance training,; Down syndrome,; Hippotherapy
MeSH Terms: conditions — Down Syndrome | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Intervention Model Description: it will be randomized controlled trial which is non probability sampling will be used. two groups of 6-14 years age will be performed in which participants will be randomly divided.group a will recieve hippotherapy and group b will recieve balance training.
Who Masked: Participant
Masking Description: participant will get seperate treatment protocols and possible effort will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hippotherapy (Experimental): Group A includes Hippo Therapy. A hippotherapy simulator is a horse riding simulator exercise machine, mimicking a horse's gait and recreating the horseback riding experience within the safety of a therapy clinic. Child with down syndrome will be seated on the stimulator for 10-15 minutes every session. The patient's pelvis moves softly, rhythmically, and repetitively when riding this action is comparable to what the human pelvis does when walking normally
  Interventions: Other: hippotherapy
- balance training (Active Comparator): The therapist modified the railing height to suit each child, ensuring the children were standing erect on the treadmill. Treadmill training completed under three conditions in 1-min training cycles. For 15 s of each minute the child could hold on to the railings with both hands, for the next 15 s with one hand, and finally with no hands on the handrails for 30 s. Each child repeated this procedure 20 Times and cool down for 5 minutes
  Interventions: Other: balance training

INTERVENTIONS:
Other: hippotherapy — A hippotherapy simulator is a horse riding simulator exercise machine, mimicking a horse's gait and recreating the horseback riding experience within the safety of a therapy clinic. Child with down syndrome will be seated on the stimulator for 10-15 minutes every session. The patient's pelvis moves softly, rhythmically, and repetitively when riding this action is comparable to what the human pelvis does when walking normally
  Arms: hippotherapy
Other: balance training — The therapist modified the railing height to suit each child, ensuring the children were standing erect on the treadmill. Treadmill training completed under three conditions in 1-min training cycles. For 15 s of each minute the child could hold on to the railings with both hands, for the next 15 s with one hand, and finally with no hands on the handrails for 30 s. Each child repeated this procedure 20 Times and cool down for 5 minutes
  Arms: balance training

SUMMARY:
Down Syndrome is a genetic condition caused by having an extra copy of chromosome 21 and 47 chromosomes instead of 46. A complete or partial extra copy of chromosome 21 is responsible for the anomaly and related structural and functional abnormalities of the body systems. Depending on the degree of abnormality, Down Syndrome has different impacts on different people as a result, differences exist in personality, abilities, talents, and physical and mental development. According to this syndrome the patients shared characteristics with one another that suggested they were siblings, including a broad, flat face, a small nose, a thick tongue, narrow palpebral fissures, obliquely positioned eyes, roundish and laterally extended cheeks, a long tongue, and varying degrees of intellectual impairment.

Prior to the study, all participants will be informed of the purpose and method of conducting the research. Each of them will sign an informed consent release to participate in the project and to process personal data for scientific purposes. This study aimed to determine the effects of hippo therapy versus balance training on balance and functional mobility in children with Down's Syndrome. Randomized clinical trials will be done. The study will be conducted in special school of education, Sargodha and Najeeb ullah rehabilitation centre, Sargodha in 10 months duration after approval of synopsis. Evaluation will be done by using pediatric balance scale, times up to go test, Functional independence measure for children, Tug test for functional mobility. Non-probability convenient sampling will be used and the subjects will be allocated to two groups by random allocation through lottery method; group A will be receiving hippo therapy and group B will be receiving balance training. Both groups will receive 8 sessions for the period of 4 weeks. Measurements of all the outcome variables will be taken at baseline, 2nd and 4th week. Data will be analyzed using SPSS-21.

DETAILED DESCRIPTION:
GROUP A:

Group A includes Hippo Therapy. A hippotherapy simulator is a horse riding simulator exercise machine, mimicking a horse's gait and recreating the horseback riding experience within the safety of a therapy clinic. Child with down syndrome will be seated on the stimulator for 10-15 minutes every session. The patient's pelvis moves softly, rhythmically, and repetitively when riding this action is comparable to what the human pelvis does when walking normally

GROUP B Group B includes balance training. The therapist modified the railing height to suit each child, ensuring the children were standing erect on the treadmill. Treadmill training completed under three conditions in 1-min training cycles. For 15 s of each minute the child could hold on to the railings with both hands, for the next 15 s with one hand, and finally with no hands on the handrails for 30 s. Each child repeated this procedure 20 Times and cool down for 5 minutes

ELIGIBILITY:
Inclusion Criteria:

* Age group of 6-14 years
* Both genders

Exclusion Criteria:

* Children with fixed deformity in LE
* Child with visual and hearing problems
* History of epilepsy

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
PEDIATRIC BALANCE SCALE | 4 weeks
  It is modified berg scale the 14 items on the scale are: standing balance, sitting balance, transfers, stepping, reaching forward with outstretched arm, reaching the floor, turning, and placing foot on stool
TIMES UP TO GO TEST | 4 weeks
  The TUG was performed from a chair 40 cm high. Participants were instructed to stand and walk 3 m to a designated area at a regular pace, then turn and return to the starting position, with the time to finish being recorded. Each participant received two trials, with the best time noted.
FUNCTIONAL INDEPENDENCE MEASURE | 4 weeks
  The maximum score on each of the 18 elements in the FIM is 7, the minimum score is 1, and the maximum possible score is 126 points. The 18 items in the FIM can be split down into two categories: five items for assessing cognitive ADL (which includes two items for communication and three items for social cognition) and thirteen items for testing motor ADL

CONTACTS AND LOCATIONS:
Overall Officials: faiza khalid, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baburamani AA, Patkee PA, Arichi T, Rutherford MA. New approaches to studying early brain development in Down syndrome. Dev Med Child Neurol. 2019 Aug;61(8):867-879. doi: 10.1111/dmcn.14260. Epub 2019 May 17. PMID 31102269